CLINICAL TRIAL: NCT04747548
Title: Supplementing Evidence-based Commercial Weight Management Program With Inhibitory Control Training in Youth: A Pilot Study
Brief Title: Inhibitory Control and Pediatric Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor, Department of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001223
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kurbo Only (Active Comparator): Participants will receive 1-month access to the Kurbo digital program.
  Interventions: Behavioral: Kurbo Only
- Kurbo + PolyRules! (Experimental): Participants will receive 1-month access to the Kurbo digital program and the PolyRules! app.
  Interventions: Behavioral: Kurbo + PolyRules!

INTERVENTIONS:
Behavioral: Kurbo Only — Kurbo is a structured behavioral weight management program for youth that focuses on diet, physical activity and mindset skills and is based on the traffic light diet developed at Stanford University. The dietary approach is based on creating an energy deficit diet to produce weight loss while also being attentive to the quality of the calories consumed. Foods are categorized into the colors of a traffic light signal based on their nutritional and caloric content, such that youth are encouraged to eat more of green and yellow foods, and less of red foods. Participants will log their daily food intake and self-monitor dietary and physical activity behaviors, incorporating behavior substitution and habit formation. Participants will also have 15 minute weekly individualized coaching sessions.
  Arms: Kurbo Only
Behavioral: Kurbo + PolyRules! — In addition to Kurbo, participants will be asked to engage in daily cognitive training using the PolyRules! app for three months. They will be instructed to start with 20-min of daily cognitive training and to progressively increase their training time to 30-min.
  Arms: Kurbo + PolyRules!

SUMMARY:
The purpose of this pilot study is to explore the benefits of supplementing the Kurbo online program with a cognitive training game (PolyRules!) among youth ages 7-13 with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Between 7-13 years old at time of enrollment
* Are able to read, write and speak English
* BMI%ile ≥ 85%ile

Exclusion Criteria:

* Concurrently enrolled in another weight loss intervention, are currently taking anti-obesity medications, or are undergoing bariatric surgery
* Have type 1 or type 2 diabetes
* Have severe cognitive delays
* Have visual/hearing impairments

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Change in BMI from baseline to 3 months to yield effect size. | Baseline, 1 month
  BMI will be calculated by aggregating participants' self-reported height in meters and weight in kilograms at baseline and at 3 months. Throughout the study, participants will be asked to self-report their weight through the Kurbo online app. This data will be used to calculate change in BMI.

SECONDARY OUTCOMES:
Improvement in self-reported diet based on adherence to dietary guidelines. | Baseline, 1 month
  Diet quality will be assessed using participant's self-reported food intake through the Kurbo online app. This data will be leveraged to assess changes in adherence to dietary guidelines for fruits and vegetables, servings of whole grains, red/processed meats and food/beverages with added sugars.
Improvement in self-reported physical activity based on adherence to physical activity guidelines. | Baseline, 1 month
  Physical activity will be assessed using participant's self-reported physical activity levels through the Kurbo online app. This data will be leveraged to assess changes in engagement in energy balance behaviors by capturing information on the type, duration and intensity of activity.
Change in performance on the cancellation task. | Baseline, 1 month
  Attention and inhibitory control will be assessed using participant's change in performance on the cancellation task. Performance will be measured by summing up the total number of errors committed within a specific time frame, such that lower scores are more favorable.
Change in performance on the countermanding task. | Baseline, 1 month
  Attention and inhibitory control will also be assessed using participant's change in performance on the countermanding task. Performance will be measured by summing the number of accurate responses within a 15 second timeframe, such that higher scores are more favorable.
Change in performance on the N-back task. | Baseline, 1 month
  Change in working memory will be assessed using participant's performance on the N-back task. Performance will be measured by looking at the number of errors such that more errors is a worse outcome.
Change in performance on the letter-number task. | Baseline, 1 month
  Change in working memory will also be assessed using participant's performance on the letter-number task. Performance will be measured by looking at error rates, such that higher error rates are worse outcomes.
Change in visuo-spatial working memory based on performance on the Corsi task. | Baseline, 1 month
  Change in visuo-spatial working memory will be assessed by participant's performance on the Corsi tasks. Performance will be measured by assessing the number of correct sequences, such that a larger number of correct sequences is a more favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah-Jeanne Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No